CLINICAL TRIAL: NCT00699751
Title: A Double-blind, Randomised, Multiple Dose, Phase III, Multicentre Study of Alpharadin in the Treatment of Patients With Symptomatic Hormone Refractory Prostate Cancer With Skeletal Metastases
Brief Title: A Phase III Study of Radium-223 Dichloride in Patients With Symptomatic Hormone Refractory Prostate Cancer With Skeletal Metastases
Acronym: ALSYMPCA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15245; BC1-06 (Other: Algeta ASA); 2007-006195-11 (EudraCT Number)
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-04

CONDITIONS: Hormone Refractory Prostate Cancer; Bone Metastases
Keywords: Hormone Refractory Prostate Cancer; Bone Metastases; Radium-223
MeSH Terms: interventions — radium Ra 223 dichloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radium-223 dichloride (Xofigo, BAY88-8223) (Experimental): Participants received radium-223 50 kilo Becquerel (kBq)/kg body weight (b.w.) for 6 intravenous (IV) administrations separated by 4 weeks intervals plus Best Standard of Care (BSoC).
  Interventions: Drug: Radium-223 dichloride (Xofigo, BAY88-8223); Drug: Best standard of care (BSoC)
- Placebo (Placebo Comparator): Participants received isotonic saline for 6 IV administrations separated by 4 weeks intervals plus Best Standard of Care (BSoC).
  Interventions: Drug: Placebo; Drug: Best standard of care (BSoC)

INTERVENTIONS:
Drug: Radium-223 dichloride (Xofigo, BAY88-8223) — Radium-223 dichloride 50 kBq/kg b.w., 6 IV administrations separated by 4 weeks intervals.
  Other Names: Alpharadin
  Arms: Radium-223 dichloride (Xofigo, BAY88-8223)
Drug: Placebo — Isotonic saline 6 IV administrations separated by 4 weeks intervals.
  Arms: Placebo
Drug: Best standard of care (BSoC) — Best standard of care is regarded as the routine standard of care at each center, for example local EBRT (External Beam Radiation Therapy), corticosteroids, antiandrogens, estrogens (e.g., stilboestrol), estramustine or ketoconazole.

SUMMARY:
ALSYMPCA (ALpharadin in SYMPtomatic Prostate CAncer) is an international Phase III clinical study to evaluate the efficacy and safety of Radium-223 dichloride in patients with hormone refractory prostate cancer and skeletal metastases.

DETAILED DESCRIPTION:
The aim of the study was to compare, in patients with symptomatic hormone refractory prostate cancer (HRPC) and skeletal metastases, the efficacy of best standard of care plus Radium-223 dichloride versus best standard of care plus placebo, with the primary efficacy endpoint being overall survival (OS).

Patients were randomised in a 2:1 allocation ratio (Radium-223 dichloride:Placebo). The study treatment consisted of 6 intravenous administrations of Radium-223 dichloride or placebo (saline) each separated by an interval of 4 weeks. The patient were followed until 3 years after first study drug administration.

Within the U.S., the trial was conducted under an IND sponsored by Bayer HealthCare Pharmaceuticals.

All patients received BSoC (Best Standard of Care).

This study has the original PCD as 14 October 2010, when a total of 316 deaths had been observed; this resulted in the Independent Data Monitoring Committee's (IDMC's) recommendation to stop the study as the primary efficacy analysis of overall survival had crossed the pre-specified boundary for efficacy. Later an updated analysis of primary endpoint in the first addendum was done with cut-off of 15 July 2011.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the prostate
* Known hormone refractory disease
* Multiple skeletal metastases (≥ 2 hot spots) on bone scintigraphy
* No intention to use cytotoxic chemotherapy within the next 6 months
* Either regular (not occasional) analgesic medication use for cancer related bone pain or treatment with EBRT (External Beam Radiation Therapy) for bone pain

Exclusion Criteria:

* Treatment with an investigational drug within previous 4 weeks, or planned during the treatment period
* Eligible for first course of docetaxel, i.e. patients who are fit enough, willing and where docetaxel is available
* Treatment with cytotoxic chemotherapy within previous 4 weeks, or planned during the treatment period, or failure to recover from adverse events due to cytotoxic chemotherapy administered more than 4 weeks ago
* Systemic radiotherapy with strontium-89, samarium-153, rhenium-186 or rhenium-188 for the treatment of bony metastases within previous 24 weeks
* Other malignancy treated within the last 5 years (except non-melanoma skin cancer or low-grade superficial bladder cancer)
* History of visceral metastasis, or visceral metastases as assessed by abdominal/pelvic CT or chest x-ray within previous 8 weeks

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 921 (Actual)
Dates: Start 2008-06; Primary Completion 2011-07 (Actual); Study Completion 2014-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Parker, MD, Study Chair — The Royal Marsden Hospital, UK
Locations (126):
- United States (7):
  - Los Angeles, California
  - Roseville, California
  - Tampa, Florida
  - New Orleans, Louisiana
  - St Louis, Missouri
  - Las Vegas, Nevada
  - Philadelphia, Pennsylvania
- Australia (12):
  - Liverpool, New South Wales
  - Randwick, New South Wales
  - St Leonards, New South Wales
  - Sydney, New South Wales
  - Wahroonga, New South Wales
  - Wollongong, New South Wales
  - Brisbane, Queensland
  - Toowoomba, Queensland
  - Adelaide, South Australia
  - Hobart, Tasmania
  - Fitzroy, Victoria
  - Nedlands, Western Australia
- Belgium (2):
  - Kortrijk
  - Ottignies
- Brazil (8):
  - Salvador, Estado de Bahia
  - Belo Horizonte, Minas Gerais
  - Rio de Janeiro, Rio de Janeiro
  - Porto Alegre, Rio Grande do Sul
  - Barretos, São Paulo
  - Piracicaba, São Paulo
  - São Paulo, São Paulo
  - Belo Horizonte
- Canada (4):
  - Edmonton, Alberta
  - London, Ontario
  - Ottawa, Ontario
  - Toronto, Ontario
- Czechia (7):
  - Brno
  - Chomutov
  - Olomouc
  - Ostrava
  - Plzen - Bory
  - Prague
  - Ústí nad Labem
- France (3):
  - La Roche-sur-Yon
  - Montbéliard
  - Saint-Cloud
- Germany (9):
  - Ulm, Baden-Wurttemberg
  - Hamburg, Hamburg
  - Frankfurt am Main, Hesse
  - Marburg, Hesse
  - Göttingen, Lower Saxony
  - Hanover, Lower Saxony
  - Dortmund, North Rhine-Westphalia
  - Mainz, Rhineland-Palatinate
  - Berlin, State of Berlin
- Hong Kong (3):
  - Chai Wan
  - Hong Kong
  - Kowloon
- Israel (4):
  - Zrifin, Israel
  - Beersheba
  - Kfar Saba
  - Tel Aviv
- Italy (5):
  - Meldola, Forlì
  - Candiolo, Torino
  - Bergamo
  - Milan
  - Reggio Emilia
- Netherlands (3):
  - Alkmaar
  - Nijmegen
  - Rotterdam
- Norway (7):
  - Ålesund
  - Bergen
  - Bodø
  - Kristiansand
  - Oslo
  - Tromsø
  - Trondheim
- Poland (7):
  - Bydgoszcz
  - Gliwice
  - Kielce
  - Krakow
  - Luiblin
  - Warsaw
  - Wroclaw
- Singapore, Singapore
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Martin
  - Prešov
  - Trnava
- Spain (8):
  - Santiago de Compostela, A Coruña
  - Barcelona, Barcelona
  - Córdoba, Córdoba
  - Alcorcón, Madrid
  - Pamplona, Pamplona
  - Valencia, Valencia
  - Barakaldo, Vizcaya
  - Zaragoza, Zaragoza
- Sweden (8):
  - Gothenburg
  - Jönköping
  - Kalmar
  - Malmo
  - Sandviken
  - Stockholm
  - Sundsvall
  - Umeå
- United Kingdom (23):
  - Bristol, Bristol
  - Romford, Essex
  - Leicester, Leicestershire
  - Manchester, Manchester
  - Bebington, Merseyside
  - Nottingham, Nottinghamshire
  - Taunton, Somerset
  - Ipswich, Suffolk
  - Guildford, Surrey
  - Sutton, Surrey
  - Coventry, Warwickshire
  - Birmingham, West Midlands
  - Belfast
  - Brighton
  - Cardiff
  - Derby
  - Hull
  - Leeds
  - Northwood
  - Plymouth
  - Sheffield
  - Southampton
  - Wolverhampton

REFERENCES:
- [Result] Parker C, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Seke M, Widmark A, Johannessen DC, Hoskin P, Bottomley D, James ND, Solberg A, Syndikus I, Kliment J, Wedel S, Boehmer S, Dall'Oglio M, Franzen L, Coleman R, Vogelzang NJ, O'Bryan-Tear CG, Staudacher K, Garcia-Vargas J, Shan M, Bruland OS, Sartor O; ALSYMPCA Investigators. Alpha emitter radium-223 and survival in metastatic prostate cancer. N Engl J Med. 2013 Jul 18;369(3):213-23. doi: 10.1056/NEJMoa1213755. PMID 23863050
- [Result] Hoskin P, Sartor O, O'Sullivan JM, Johannessen DC, Helle SI, Logue J, Bottomley D, Nilsson S, Vogelzang NJ, Fang F, Wahba M, Aksnes AK, Parker C. Efficacy and safety of radium-223 dichloride in patients with castration-resistant prostate cancer and symptomatic bone metastases, with or without previous docetaxel use: a prespecified subgroup analysis from the randomised, double-blind, phase 3 ALSYMPCA trial. Lancet Oncol. 2014 Nov;15(12):1397-406. doi: 10.1016/S1470-2045(14)70474-7. Epub 2014 Oct 17. PMID 25439694
- [Result] Sartor O, Coleman R, Nilsson S, Heinrich D, Helle SI, O'Sullivan JM, Fossa SD, Chodacki A, Wiechno P, Logue J, Widmark A, Johannessen DC, Hoskin P, James ND, Solberg A, Syndikus I, Vogelzang NJ, O'Bryan-Tear CG, Shan M, Bruland OS, Parker C. Effect of radium-223 dichloride on symptomatic skeletal events in patients with castration-resistant prostate cancer and bone metastases: results from a phase 3, double-blind, randomised trial. Lancet Oncol. 2014 Jun;15(7):738-46. doi: 10.1016/S1470-2045(14)70183-4. Epub 2014 May 13. PMID 24836273
- [Result] Delacruz A, Arauz G, Curley T, Lindo A, Jensen T. Nursing management of patients with castration-resistant prostate cancer undergoing radium-223 dichloride treatment. Clin J Oncol Nurs. 2015 Apr;19(2):E31-5. doi: 10.1188/15.CJON.E31-E35. PMID 25840395
- [Result] Humm JL, Sartor O, Parker C, Bruland OS, Macklis R. Radium-223 in the treatment of osteoblastic metastases: a critical clinical review. Int J Radiat Oncol Biol Phys. 2015 Apr 1;91(5):898-906. doi: 10.1016/j.ijrobp.2014.12.061. PMID 25832684
- [Result] Nilsson S. Alpha-emitter radium-223 in the management of solid tumors: current status and future directions. Am Soc Clin Oncol Educ Book. 2014:e132-9. doi: 10.14694/EdBook_AM.2014.34.e132. PMID 24857093
- [Result] Den RB, Doyle LA, Knudsen KE. Practical guide to the use of radium 223 dichloride. Can J Urol. 2014 Apr;21(2 Supp 1):70-6. PMID 24775727
- [Result] Shirley M, McCormack PL. Radium-223 dichloride: a review of its use in patients with castration-resistant prostate cancer with symptomatic bone metastases. Drugs. 2014 Apr;74(5):579-86. doi: 10.1007/s40265-014-0198-4. PMID 24610703
- [Result] Wissing MD, van Leeuwen FW, van der Pluijm G, Gelderblom H. Radium-223 chloride: Extending life in prostate cancer patients by treating bone metastases. Clin Cancer Res. 2013 Nov 1;19(21):5822-7. doi: 10.1158/1078-0432.CCR-13-1896. Epub 2013 Sep 19. PMID 24052017
- [Result] Joung JY, Ha YS, Kim IY. Radium Ra 223 dichloride in castration-resistant prostate cancer. Drugs Today (Barc). 2013 Aug;49(8):483-90. doi: 10.1358/dot.2013.49.8.1968670. PMID 23977665
- [Derived] Parker C, Zhan L, Cislo P, Reuning-Scherer J, Vogelzang NJ, Nilsson S, Sartor O, O'Sullivan JM, Coleman RE. Effect of radium-223 dichloride (Ra-223) on hospitalisation: An analysis from the phase 3 randomised Alpharadin in Symptomatic Prostate Cancer Patients (ALSYMPCA) trial. Eur J Cancer. 2017 Jan;71:1-6. doi: 10.1016/j.ejca.2016.10.020. Epub 2016 Dec 6. PMID 27930924
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe. — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with progressive symptomatic hormone refractory prostate cancer (HRPC), with at least 2 skeletal metastases on bone scan and no known visceral metastases, could participate in the study.
Pre-assignment Details: Subjects were to be randomized in a 2:1, a total of 921 subjects were enrolled in the study and were randomized to receive either Alpharadin [Radium-223 dichloride (Xofigo, BAY88-8223)] or placebo study treatment, which resulted in 614 subjects enrolled in the Alpharadin group and 307 enrolled in the placebo group.
Groups:
- Radium-223 Dichloride (Xofigo, BAY88-8223): Participants received BSoC plus radium223 50 kBq/kg body weight for 6 IV administrations separated by 4 weeks intervals.
- Placebo: Participants received BSoC plus isotonic saline for 6 IV administrations separated by 4 weeks intervals in double-blind phase; Participants received radium223 50 kBq/kg body weight for 6 intravenous administrations separated by 4 weeks intervals after unblinding to the end of study.
Period: Period 1: Without/Before Drug Switch
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Started | 614 | 307
Participants Received Treatment | 600 | 301
Entered 3-Year Follow-up Period | 407 (Participants were not required to complete all 6 injections to enter to 3-year follow-up period.) | 168 (Participants were not required to complete all 6 injections to enter to 3-year follow-up period.)
Completed 3-Year Follow-up Period | 49 | 12
Completed | 389 (Completed all 6 injections) | 145 (Completed all 6 injections)
Not Completed | 225 | 162
Not completed — Investigator Request | 27 | 27
Not completed — Death | 28 | 29
Not completed — Subject Request | 43 | 23
Not completed — Other | 30 | 20
Not completed — Adverse Event | 97 | 63
Period: Period 2:Switched From Placebo to Xofigo
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Started | 0 | 26 (Participants in the placebo group switched to Xofigo treatment)
Participants Received Treatment | 0 | 24
Entered 3-Year Follow-up Period | 0 | 15
Completed 3-Year Follow-up Period | 0 | 0
Completed | 0 | 17 (Completed all 6 injections)
Not Completed | 0 | 9
Not completed — Adverse Event | 0 | 4
Not completed — Investigator Request | 0 | 1
Not completed — Completion page not expected | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Radium-223 Dichloride (Xofigo, BAY88-8223): Radium-223 50 kilo Becquerel (kBq)/kg body weight (b.w.) for 6 intravenous (IV) administrations separated by 4 weeks intervals plus BSoC.
- Placebo: Isotonic saline for 6 IV administrations separated by 4 weeks intervals plus BSoC.
- Total: Total of all reporting groups
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo | Total
Number analyzed (Participants) | 614 | 307 | 921
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.2 (8.10) | 70.8 (7.87) | 70.4 (8.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 614 | 307 | 921
Total Alkaline Phosphatase (ALP) [Number; unit: Participants] — The total amount of ALP in the blood was determined at baseline.
  Participants
    < 220 U/L | 348 | 169 | 517
    ≥ 220 U/L | 266 | 138 | 404
Current use of bisphosphonates [Number; unit: Participants] — Subjects may have been on bisphosphonate therapy during the study.
  Participants
    Yes | 250 | 124 | 374
    No | 364 | 183 | 547
Any prior use of docetaxel [Number; unit: Participants]
  Yes | 352 | 174 | 526
  No | 262 | 133 | 395

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival was defined as the time from date of randomization to the date of death.
Time Frame: From randomization to death due to any cause until approximately 3 years after start of enrollment, the data was collected up to the second data analysis date (15 JUL 2011)
Population: The intent-to-treat (ITT) population was defined as all randomized subjects.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | 14.9 [13.9 to 16.1] | 11.3 [10.1 to 12.8]
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of overall survival, and also for the secondary endpoints, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.00005, Log Rank; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.691, 95% CI 2-sided [0.578 to 0.827] — The hazard ratio (Alpharadin:Placebo) is from a Cox proportional hazards model stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel

2. Secondary Outcome: Time to Total Alkaline Phosphatase (ALP) Progression
Description: The time from the first study drug administration to when ALP progression was observed, defined as: 1) In subjects with no ALP decline from baseline; a greater than or equal to 25% increase from baseline value and an increase in absolute value of greater than or equal to 2 ng/mL, at least 12 weeks from baseline; 2) In subjects with initial ALP decline from baseline; the time from start of treatment to first ALP increase that is greater than or equal to 25% increase and at least 2 ng/mL above the nadir value, which was confirmed by a second value obtained 3 or more weeks later
Time Frame: From randomization to first ALP progression until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | 7.4 [7.1 to NA] — 95% Confidence Interval upper limit is not estimable due to insufficient number of participants with events. | 3.8 [3.6 to 4.2]
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of time to total ALP progression, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.00001, Log Rank; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.169, 95% CI 2-sided [0.131 to 0.22] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percentage of Participants With Total ALP Response at Week 12
Description: ALP levels were measured in participants' blood at Week 12 and compared to baseline values. A confirmed total ALP response (either >/= 30% or 50% reduction from baseline) was confirmed by a second total ALP value approximately 4 weeks later.
Time Frame: At Baseline and Week 12
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 497 | 211
Percentage of participants
  >=30% reduction of ALP in blood level | 59.4 | 6.2
  >=50% reduction of ALP in blood level | 32.6 | 1.4
  Confirmed Total ALP Response (>=30%) | 47.1 | 3.3
  Confirmed Total ALP Response (>=50%) | 27.4 | 0.9
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of >=30% reduction in blood level, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — >=30% reduction in blood level; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 2: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of >=50% reduction in blood level, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — >=50% reduction in blood level; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 3: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Confirmed Total ALP Response (>=30%), is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Confirmed Total ALP Response (>=30%); adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 4: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Confirmed Total ALP Response (>=50%), is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Confirmed Total ALP Response (>=50%); adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

4. Secondary Outcome: Percentage of Participants With Total ALP Response at End of Treatment (EOT; Week 24 or at the Time the Patient Dies or Discontinues Treatment Phase)
Description: ALP levels were measured in participants' blood at EOT (Week 24) and compared to baseline values. A confirmed total ALP response (>/=50% reduction from baseline) was confirmed by a second total ALP value approximately 4 weeks later.
Time Frame: At Baseline and End of Treatment (Week 24 or at the time the patient dies or discontinues treatment phase)
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 589 | 288
Percentage of participants
  >=30% reduction of ALP in blood level | 59.9 | 4.5
  >=50% reduction of ALP in blood level | 34.6 | 1.7
  Confirmed Total ALP Response (>=50%) | 13.9 | 1
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — >=30% reduction in blood level; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 2: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — >=50% reduction in blood level; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 3: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Confirmed Total ALP Response (>=50%); adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

5. Secondary Outcome: Percentage of Participants With Total ALP Normalization at Week 12
Description: The return of total ALP value to within normal range at 12 weeks in 2 consecutive measurements (at least 2 weeks apart) after start of treatment in subjects who had ALP above the upper limit of normal (ULN) at baseline.
Time Frame: At Baseline and Week 12
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 321 | 140
Percentage of participants | 34 | 1.4
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Total ALP normalization, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — Total ALP normalization; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

6. Secondary Outcome: Percentage Change From Baseline in Total ALP at Week 12
Description: ALP level was measured in subject's blood at Week 12 and the percent change from the baseline value was calculated (ALP level at week 12 minus ALP level at baseline)/(ALP level at baseline)*100
Time Frame: At Baseline and Week 12
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 497 | 211
Percentage change | -32.2 (1.80) | 37.2 (2.77)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Percentage change from baseline, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, ANCOVA — Percentage Change from Baseline; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

7. Secondary Outcome: Maximum Percentage Decrease From Baseline in Total ALP up to Week 12
Description: ALP level was measured in participant's blood up to week 12 and the maximum percent decrease from the baseline up to Week 12 value was calculated as the minimum value of [(ALP level up to week 12 minus ALP level at baseline)/(ALP level at baseline)*100] by participant, and set to zero if no decrease from baseline.
Time Frame: From baseline to Week 12
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 582 | 284
Percentage change | -38.9 (0.76) | -5.9 (1.09)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Maximum Percentage decrease from baseline to week 12, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, ANCOVA — Maximum Percentage decrease from baseline to week 12; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

8. Secondary Outcome: Percentage Change From Baseline in Total ALP at EOT (Week 24 or at the Time the Patient Dies or Discontinues Treatment Phase)
Description: ALP level was measured in subject's blood at EOT (Week 24) and the percent change from the baseline value was calculated (ALP level at EOT minus ALP level at baseline)/(ALP level at baseline)*100
Time Frame: At Baseline and End of Treatment (Week 24 or at the time the patient dies or discontinues treatment phase)
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 589 | 288
Percent change | -29.9 (3.13) | 62.1 (4.48)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p < 0.001, ANCOVA — Percentage change from baseline; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

9. Secondary Outcome: Maximum Percentage Decrease From Baseline in Total ALP During the 24 Week Treatment
Description: ALP level was measured in participant's blood during the 24 week treatment (up to EOT) and the maximum percent decrease from baseline during the 24 week treatment value was calculated as the minimum value of [(ALP level up to week 24 minus ALP level at baseline)/(ALP level at baseline)*100] by participant, and set to zero if no decrease from baseline.
Time Frame: From baseline During the 24 Week Treatment
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 589 | 288
Percentage change | -44.4 (0.80) | -7.5 (1.14)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Maximum Percentage decrease from baseline during the 24 week treatment, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, ANCOVA — Maximum Percentage decrease from baseline during the 24 week treatment; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

10. Secondary Outcome: Time to Prostate Specific Antigen (PSA) Progression
Description: The time from the first study drug administration to when PSA progression was observed, defined as: 1) In subjects with no PSA decline from baseline; a greater than or equal to 25% increase from baseline value and an increase in absolute value of greater than or equal to 2 ng/mL, at least 12 weeks from baseline; 2) In subjects with initial PSA decline from baseline; the time from start of treatment to first PSA increase that is greater than or equal to 25% increase and at least 2 ng/mL above the nadir value, which was confirmed by a second value obtained 3 or more weeks later
Time Frame: From randomization to first PSA progression until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | 3.6 [3.5 to 3.8] | 3.4 [3.3 to 3.5]
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Time to PSA progression, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.00001, Log Rank — Time to Prostate Specific Antigen (PSA) progression; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.643, 95% CI 2-sided [0.539 to 0.768] — [estimate comment as in outcome 1, analysis 1]

11. Secondary Outcome: Percentage of Participants With PSA Response at Week 12
Description: PSA levels were measured in participants' blood at Week 12 and compared to baseline values. A confirmed PSA response (>/=50% reduction from baseline) was confirmed by a second PSA value approximately 4 weeks later.
Time Frame: At Baseline and Week 12
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 493 | 210
Percentage of participants
  >=30% reduction of PSA in blood level | 16.4 | 6.2
  >=50% reduction of PSA in blood level | 7.7 | 4.3
  Confirmed PSA Response (>=50%) | 5.7 | 1.9
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — >=30% reduction in blood level; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 2: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.106, Cochran-Mantel-Haenszel — >=50% reduction in blood level; adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 3: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Confirmed PSA Response(>=50%), is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.032, Cochran-Mantel-Haenszel — Confirmed PSA Response(>=50%); Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

12. Secondary Outcome: Percentage of Participants With PSA Response at EOT (Week 24 or at the Time the Patient Dies or Discontinues Treatment Phase)
Description: PSA levels were measured in participants' blood at EOT (Week 24) and compared to baseline values. A confirmed PSA response (>/=50% reduction from baseline) was confirmed by a second PSA value approximately 4 weeks later.
Time Frame: At Baseline and End of Treatment (Week 24 or at the time the patient dies or discontinues treatment phase)
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Number; unit: Percentage of participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 590 | 286
Percentage of participants
  >=30% reduction in blood level | 14.2 | 4.5
  >=50% reduction in blood level | 9 | 3.1
  Confirmed PSA Response (>=50%) | 6.1 | 1.7
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel — >=30% reduction in blood level; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 2: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.002, Cochran-Mantel-Haenszel — >=50% reduction in blood level; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel
Statistical Analysis 3: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; [analysis description as in outcome 11, analysis 3]; Test type: Superiority or Other; p = 0.005, Cochran-Mantel-Haenszel — Confirmed PSA Response(>=50%); Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

13. Secondary Outcome: Percentage Change From Baseline in PSA at Week 12
Description: PSA level was measured in subject's blood at Week 12 and the percent change from the baseline value was calculated (PSA level at week 12 minus PSA level at baseline)/(PSA level at baseline)*100
Time Frame: At Baseline and Week 12
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 493 | 210
Percent change | 83.3 (152.48) | 543.8 (233.69)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Percentage change from baseline in PSA at Week 12, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.160, ANCOVA — Percentage change from baseline in PSA at Week 12; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

14. Secondary Outcome: Maximum Percentage Decrease From Baseline in PSA up to Week 12
Description: PSA level was measured in participant's blood up to Week 12 and the maximum percent decrease from the baseline up to week 12 value was calculated as the minimum value of [(PSA level up to week 12 minus PSA level at baseline)/(PSA level at baseline)*100] by participant, and set to zero if no decrease from baseline.
Time Frame: From baseline up to Week 12
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 581 | 283
Percentage change | -13.0 (0.90) | -7.8 (1.28)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Maximum Percentage Decrease from Baseline up to Week 12, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.004, ANCOVA — Maximum Percentage Decrease from Baseline up to Week 12; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

15. Secondary Outcome: Percentage Change From Baseline in PSA at EOT (Week 24 or at the Time the Patient Dies or Discontinues Treatment Phase)
Description: PSA level was measured in subject's blood at EOT (Week 24) and the percent change from the baseline value was calculated (PSA level at EOT minus PSA level at baseline)/(PSA level at baseline)*100
Time Frame: At Baseline and End of Treatment (Week 24 or at the time the patient dies or discontinues treatment phase)
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 590 | 286
Percentage change | 144.3 (15.38) | 191.1 (22.1)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Percentage change from baseline in PSA at EOT, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.009, ANCOVA — Percentage change from baseline in PSA at EOT; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

16. Secondary Outcome: Maximum Percentage Decrease From Baseline in PSA Response During the 24 Week Treatment Period
Description: PSA level was measured in participant's blood during the 24 week treatment (up to EOT) and the maximum percent decrease from baseline during the 24 Week treatment value was calculated as the minimum value of [(PSA level up to week 24 minus PSA level at baseline)/(PSA level at baseline)*100] by participant, and set to zero if no decrease from baseline.
Time Frame: From baseline to End of Treatment (Week 24; 4 weeks post last injection)
Population: Participants in The ITT population and had no missing values for this outcome measure
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 590 | 286
Percentage change | -16.4 (1.01) | -9.3 (1.45)
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Maximum Percentage Decrease from Baseline in PSA response During the 24 Week Treatment Period, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p < 0.001, ANCOVA — Maximum Percentage Decrease from Baseline in PSA response During the 24 Week Treatment Period; Adjusting for the binary stratification factors, total ALP, current use of Bisphosphonates and prior use of Docetaxel

17. Secondary Outcome: Time to First Skeletal Related Event (SRE)
Description: A skeletal related event is the use of external beam radiotherapy to relieve skeletal symptoms or the occurrence of new symptomatic pathological bone fractures (vertebral or non-vertebral) or the occurrence of spinal cord compression or a tumour related orthopaedic surgical intervention. For all other events, the start date of the event/medication/therapy was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From randomization to first first SRE until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | 16.4 [14.3 to 18.3] | 8.1 [6.7 to 11.9]
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of time to first SRE, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.00012, Log Rank — Time to first Skeletal Related Event (SRE); Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.657, 95% CI 2-sided [0.529 to 0.814] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Time to Occurrence of First Use of External Beam Radiation Therapy (EBRT) to Relieve Skeletal Symptoms
Description: The start date of therapy was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From randomization to first EBRT until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | 18 [15.9 to 20.6] | 10.7 [7.6 to 18.5]
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of time to EBRT, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.00008, Log Rank — Time to External Beam Radiotherapy; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.639, 95% CI 2-sided [0.511 to 0.8] — [estimate comment as in outcome 1, analysis 1]

19. Secondary Outcome: Time to Occurrence of First Use of Radioisotopes to Relieve Skeletal Symptoms
Description: The start date of the radioisotopes was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From randomization to first use of radioisotopes until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | NA [NA to NA] — Median survival time is not reached | NA [NA to NA] — Median survival time is not reached
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Time to Receiving Radio-isotope, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.00191, Log Rank — stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.344, 95% CI 2-sided [0.17 to 0.695] — [estimate comment as in outcome 1, analysis 1]

20. Secondary Outcome: Time to Occurrence of First New Symptomatic Pathological Bone Fractures, Vertebral and Non-vertebral
Description: The start date of the event was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From randomization to occurrence of first new symptomatic pathological bone fractures until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | NA [NA to NA] — Median survival time is not reached. | NA [NA to NA] — Median survival time is not reached.
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Time to Pathological Bone Fracture, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.53277, Log Rank — Time to Pathological Bone Fracture; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.847, 95% CI 2-sided [0.504 to 1.426] — [estimate comment as in outcome 1, analysis 1]

21. Secondary Outcome: Time to Occurrence of First Tumor Related Orthopedic Surgical Intervention
Description: The start date of the intervention was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From randomization to occurrence of first tumor related orthopedic surgical intervention until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | NA [NA to NA] — Median survival time is not reached | NA [NA to NA] — Median survival time is not reached
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Time to Surgical Intervention, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.89567, Log Rank — Time to Surgical Intervention; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.949, 95% CI 2-sided [0.435 to 2.07] — [estimate comment as in outcome 1, analysis 1]

22. Secondary Outcome: Time to Occurrence of First Spinal Cord Compression
Description: The start date of the compression was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From randomization to first spinal cord compression until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | NA [NA to NA] — Median survival time is not reached | NA [NA to NA] — Median survival time is not reached
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Time to Spinal Cord Compression, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.14486, Log Rank — Time to Spinal Cord Compression; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.404 to 1.145] — [estimate comment as in outcome 1, analysis 1]

23. Secondary Outcome: Time to Occurrence of First Start of Any Other Anti-cancer Treatment
Description: The start date of the treatment was used as the time of the event. If an event has not occurred at the time of the analysis or the patient has been lost to follow-up, the time-to-event variables will be censored at the last disease assessment date.
Time Frame: From randomization to first start of any other anti-cancer treatment until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | 15.4 [12.6 to 17] | 12.7 [11.0 to 14.7]
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Time to Other Cancer Treatment, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.00932, Log Rank — Time to Other Cancer Treatment; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.727, 95% CI 2-sided [0.571 to 0.925] — [estimate comment as in outcome 1, analysis 1]

24. Secondary Outcome: Time to Occurrence of First Deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG PS) by at Least 2 Points From Baseline
Description: ECOG scores were: 0 = fully active; 1 = restricted in physically strenuous activity; 2 = ambulatory and capable of all self-care but unable to work; 3 = capable of only limited self-care; 4 = completely disabled; 5 = death. The visit at which a 2-point or more deterioration in PS was observed was the time of the event. ECOG was assessed at every visit. If a marked deterioration in PS has not occurred at the time of the analysis or the participant was lost to follow-up, the time-to-event variables were censored at the last assessment date.
Time Frame: From randomization to first deterioration of Eastern Cooperative Oncology Group Performance Status (ECOG PS) until approximately 3 years after start of enrollment
Population: The ITT population was all randomized subjects
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Months | 23.4 [20.4 to 26.5] | 18.4 [13.1 to 24.5]
Statistical Analysis 1: Comparison: Radium-223 Dichloride (Xofigo, BAY88-8223) vs Placebo; The null hypothesis for the comparison of Time to Marked Deterioration of ECOG PS, is that there is no difference between Alpharadin and placebo for that endpoint; the alternative hypothesis is that a difference exists; Test type: Superiority or Other; p = 0.00187, Log Rank — Time to Marked Deterioration of ECOG PS; Stratified by total ALP, current use of bisphosphonates and prior use of Docetaxel; Hazard Ratio (HR) = 0.69, 95% CI 2-sided [0.546 to 0.873] — [estimate comment as in outcome 1, analysis 1]

25. Other Pre Specified Outcome: Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) at Week 0.
Description: ECOG PS was defined as: 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature (eg, light house work, office work); 2 = Ambulatory and capable of all self-care but unable to carry out work activities. Up and about > 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair > 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair; or 5 = Dead.
Time Frame: Week 0
Population: Participants in The ITT population and with ECOG analyzed
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 600 | 305
Participants
  ECOG Grade 0 | 136 | 72
  ECOG Grade 1 | 376 | 191
  ECOG Grade 2 | 82 | 40
  ECOG Grade 3 | 6 | 1
  ECOG Grade 4 | 0 | 0
  ECOG Grade 5 | 0 | 0
  Missing | 0 | 1

26. Other Pre Specified Outcome: Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) at Week 8.
Description: as for outcome 25
Time Frame: Week 8
Population: Participants in The ITT population and with ECOG analyzed
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 569 | 267
Participants
  ECOG Grade 0 | 133 | 49
  ECOG Grade 1 | 315 | 142
  ECOG Grade 2 | 103 | 53
  ECOG Grade 3 | 13 | 15
  ECOG Grade 4 | 0 | 3
  ECOG Grade 5 | 1 | 1
  Missing | 4 | 4

27. Other Pre Specified Outcome: Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) at Week 16.
Description: as for outcome 25
Time Frame: Week 16
Population: Participants in The ITT population and with ECOG analyzed
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 471 | 196
Participants
  ECOG Grade 0 | 101 | 29
  ECOG Grade 1 | 257 | 113
  ECOG Grade 2 | 85 | 42
  ECOG Grade 3 | 19 | 11
  ECOG Grade 4 | 4 | 0
  ECOG Grade 5 | 0 | 0
  Missing | 5 | 1

28. Other Pre Specified Outcome: Number of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) at Week 24.
Description: as for outcome 25
Time Frame: Week 24
Population: Participants in The ITT population and with ECOG analyzed
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 363 | 138
Participants
  ECOG Grade 0 | 74 | 22
  ECOG Grade 1 | 181 | 66
  ECOG Grade 2 | 85 | 36
  ECOG Grade 3 | 17 | 10
  ECOG Grade 4 | 5 | 4
  ECOG Grade 5 | 0 | 0
  Missing | 1 | 0

29. Other Pre Specified Outcome: Absolute Scores for Functional Assessment of Cancer Therapy - Prostate (FACT-P) Trial Outcome Index (TOI)
Description: The FACT-P was 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being. It was supplemented by 12 questions relating to prostate cancer. The absolute score for the FACT-P TOI domain (physical and social well-being and prostate specific score) was calculated for each visit. Prostate Cancer Trial Outcome Index (TOI): Physical Well-being (PWB) + Functional Well-being (FWB) + Prostate Cancer (PCS). Score ranges from 0 (worst) to 104 (best).
Time Frame: Baseline, Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  Week 0 (Baseline) | 65.00 [17.0 to 104.0] | 64.00 [23.0 to 96.0]
  Week 16 | 65.00 [11.0 to 98.0] | 61.31 [19.0 to 96.5]
  Week 24 | 61.00 [17.0 to 102.0] | 60.00 [17.0 to 97.0]
  Follow-up Visit 2 (Week 42) | 61.00 [10.0 to 95.0] | 60.5 [16.7 to 97.0]

30. Other Pre Specified Outcome: Changes From Baseline for FACT-P Trial Outcome Index (TOI) at Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Description: The FACT-P was 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being. It was supplemented by 12 questions relating to prostate cancer. The absolute score for the FACT-P TOI domain (physical and social well-being and prostate specific score) was calculated for each visit. Possible scores were 0 to 104; the higher the score, the better the quality of life. The changes from baseline (range -104 to 104) in the domain FACT-P TOI were summarized using descriptive statistics at Week 16, Week 24, and Follow-up Visit 2.
Time Frame: Baseline, Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  At Week 16 | -1.55 [-49.3 to 38.0] | -4.15 [-43.0 to 46.0]
  At Week 24 | -4.00 [-60.4 to 40.0] | -5.67 [-39.0 to 41.0]
  At Follow-up Visit 2 (Week 42) | -5.00 [-89.0 to 44.5] | -5.5 [-47.4 to 25.0]

31. Other Pre Specified Outcome: Absolute Scores for Physical Well Being, Social/Family Well Being, Emotional Well Being, Functional Well Being, and the Prostate Cancer Subscale at Week 16
Description: The FACT-P was 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being and was supplemented by 12 questions relating to prostate cancer. Possible scores for each subscale were 0 to 28; 0 to 28; 0 to 24; 0 to 28; and 0 to 48, respectively. All FACT-P items are scored on a scale of 0-4 representing the extent to which the item reflects the experience of the individual completing the instrument (0 - Not at all; 4 - Very much). Higher scores indicate better quality of life. The absolute score of the FACT-P total score was calculated at Week 16.
Time Frame: At Week 16
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  physical well being | 20.00 [3.0 to 28.0] | 19.83 [1.0 to 28.0]
  social/family well being | 22.00 [0.0 to 28.0] | 21.50 [0.0 to 28.0]
  emotional well being | 18.0 [0.0 to 24.0] | 16.80 [2.0 to 24.0]
  functional well being | 16.0 [0.0 to 28.0] | 15.0 [0.0 to 28.0]
  the prostate cancer subscale | 29.00 [1.0 to 46.9] | 27.60 [9.0 to 42.5]

32. Other Pre Specified Outcome: Absolute Scores for Physical Well Being, Social/Family Well Being, Emotional Well Being, Functional Well Being, and the Prostate Cancer Subscale at Week 24
Description: The FACT-P was 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being and was supplemented by 12 questions relating to prostate cancer. Possible scores for each subscale were 0 to 28; 0 to 28; 0 to 24; 0 to 28; and 0 to 48, respectively. All FACT-P items are scored on a scale of 0-4 representing the extent to which the item reflects the experience of the individual completing the instrument (0 - Not at all; 4 - Very much). Higher scores indicate better quality of life. The absolute score of the FACT-P total score was calculated at Week 24.
Time Frame: At Week 24
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  physical well being | 19.00 [3.0 to 28.0] | 18.67 [3.0 to 28.0]
  social/family well being | 21.00 [0.0 to 28.0] | 21.00 [9.0 to 28.0]
  emotional well being | 17.00 [4.0 to 24.0] | 16.00 [1.2 to 24.0]
  functional well being | 15.00 [0.0 to 28.0] | 14.00 [0.0 to 28.0]
  the prostate cancer subscale | 28.00 [3.6 to 46.0] | 27.64 [5.0 to 43.0]

33. Other Pre Specified Outcome: Absolute Scores for Physical Well Being, Social/Family Well Being, Emotional Well Being, Functional Well Being, and the Prostate Cancer Subscale at Follow-up Visit 2 (Week 42)
Description: The FACT-P was 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being and was supplemented by 12 questions relating to prostate cancer. Possible scores for each subscale were 0 to 28; 0 to 28; 0 to 24; 0 to 28; and 0 to 48, respectively. All FACT-P items are scored on a scale of 0-4 representing the extent to which the item reflects the experience of the individual completing the instrument (0 - Not at all; 4 - Very much). Higher scores indicate better quality of life. The absolute score of the FACT-P total score was calculated at Follow-up Visit 2.
Time Frame: At Follow-up Visit 2 (Week 42)
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  physical well being | 19.00 [0.0 to 28.0] | 18.00 [1.0 to 28.0]
  social/family well being | 22.00 [0.0 to 28.0] | 22.00 [9.0 to 33.8]
  emotional well being | 17.00 [0.0 to 24.0] | 16.00 [3.0 to 24.0]
  functional well being | 14.00 [1.0 to 28.0] | 14.00 [4.0 to 28.0]
  the prostate cancer subscale | 28.00 [3.0 to 42.0] | 29.00 [6.5 to 43.0]

34. Other Pre Specified Outcome: Absolute Scores for FACT-P Total Score at Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Description: The FACT-P was 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being. It was supplemented by 12 questions relating to prostate cancer. The absolute score of the FACT-P total score (physical, social/family, emotional, and functional well-being and prostate specific score) was calculated at Week 16, Week 24, and Follow-up Visit 2.FACT-P Total Score: Physical Well-being (PWB) + Social/Family Well-being (SWB) + Emotional Well-being (EWB) + Functional Well-being (FWB) + Prostate Cancer (PCS). Score ranges from 0 (worst) to 156 (best).
Time Frame: At Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  At Week 16 | 100.68 [30.0 to 147.0] | 99.90 [33.7 to 144.0]
  At Week 24 | 98.00 [41.8 to 152.0] | 97.5 [47.0 to 149.0]
  At Follow-up Visit 2 (Week 42) | 97.83 [41.0 to 145.0] | 97.38 [40.9 to 147.8]

35. Other Pre Specified Outcome: Change From Baseline for FACT-P Total Score at Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Description: The FACT-P was 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being. It was supplemented by 12 questions relating to prostate cancer. Total possible score was 156; a higher score indicates a better quality of life. The changes from baseline in the FACT-P total score (physical, social/family, emotional, and functional well-being and prostate specific score) were calculated at Week 16, Week 24, and Follow-up Visit 2. Possible range was -156 to 156.
Time Frame: Baseline, Week 16, Week 24, and Follow-up Visit 2 (week 42)
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  At Week 16 | -2.00 [-58.0 to 58.0] | -5.67 [-58.0 to 47]
  At Week 24 | -5.00 [-67.2 to 63.5] | -9.40 [-42.8 to 48.8]
  At Follow-up Visit 2 (Week 42) | -6.17 [-97.0 to 63.5] | -7.00 [-54.7 to 23.7]

36. Other Pre Specified Outcome: Absolute Scores for Functional Assessment of Cancer Therapy - General (FACT-G) Total Score at Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Description: The FACT-G instrument consisted of 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being. The FACT-G absolute total score (physical, social/family, emotional, and functional well-being) was calculated at Week 16, Week 24, and Follow-up Visit 2. FACT-G Total Score: Physical Well-being (PWB) + Social/Family Well-being (SWB) + Emotional Well-being (EWB) + Functional Well-being (FWB). Score ranges from 0 (worst) to 108 (best).
Time Frame: At Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  At Week 16 | 73.00 [17.0 to 106.0] | 72.00 [27.7 to 108.0]
  At Week 24 | 71.00 [28.0 to 107.0] | 69.00 [37.0 to 106.0]
  At Follow-up Visit 2 (Week 42) | 70.00 [22.0 to 107.0] | 70.25 [32.2 to 104.8]

37. Other Pre Specified Outcome: Change From Baseline for FACT-G Total Score at Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Description: The FACT-G instrument consisted of 27 questions relating to 4 domains: physical, social/family, emotional, and functional well-being. Total possible score was 108; a higher score indicates a better quality of life. The changes from baseline in the FACT-G total score (physical, social/family, emotional, and functional well-being) were calculated at Week 16, Week 24, and Follow-up Visit 2. Possible range was -108 to 108.
Time Frame: Baseline, Week 16, Week 24, and Follow-up Visit 2 (Week 42)
Population: The ITT population was all randomized subjects
Measure: Median (Full Range); unit: Scores on a scale
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 614 | 307
Scores on a scale
  At Week 16 | -1.00 [-38.3 to 40.0] | -4.00 [-53.0 to 32.8]
  At Week 24 | -4.08 [-49.0 to 49.5] | -7.00 [-35.8 to 41.8]
  At Follow-up Visit 2 (Week 42) | -3.67 [-58.0 to 40.5] | -6.00 [-33.8 to 18.7]

38. Other Pre Specified Outcome: Number of Participants in the Euro Quality of Life (EQ-5D) Components for Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression at Week 16
Description: The EQ-5D questionnaire was given to the subject at each visit. The EQ-5D questionnaire consisted of 5 ordinal categorical responses (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Number of participants with EQ-5D at Week 16, as measured by this questionnaire, was counted. The scores for the EQ-5D dimensions are assigned according to the level of problems reported (1 'no problems'; 2 'some problems'; 3 'extreme problems').
Time Frame: Week 16
Population: The ITT population was all randomized subjects with with EQ-5D analyzed.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 477 | 205
Participants
  mobility - Grade 1 | 191 | 64
  mobility - Grade 2 | 278 | 129
  mobility - Grade 3 | 7 | 10
  mobility - Missing | 1 | 2
  self-care - Grade 1 | 346 | 140
  self-care - Grade 2 | 123 | 54
  self-care - Grade 3 | 7 | 10
  self-care - Missing | 1 | 1
  usual activities - Grade 1 | 199 | 67
  usual activities - Grade 2 | 233 | 105
  usual activities - Grade 3 | 44 | 32
  usual activities - Missing | 1 | 1
  pain/discomfort - Grade 1 | 79 | 23
  pain/discomfort - Grade 2 | 351 | 159
  pain/discomfort - Grade 3 | 46 | 22
  pain/discomfort - Missing | 1 | 1
  anxiety/depression - Grade 1 | 285 | 104
  anxiety/depression - Grade 2 | 171 | 95
  anxiety/depression - Grade 3 | 15 | 4
  anxiety/depression - Missing | 6 | 2

39. Other Pre Specified Outcome: Number of Participants in the Euro Quality of Life (EQ-5D) Components for Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression at Week 24
Description: The EQ-5D questionnaire was given to the subject at each visit. The EQ-5D questionnaire consisted of 5 ordinal categorical responses (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Number of participants with EQ-5D at Week 24, as measured by this questionnaire, was counted. The scores for the EQ-5D dimensions are assigned according to the level of problems reported (1 'no problems'; 2 'some problems'; 3 'extreme problems').
Time Frame: Week 24
Population: The ITT population was all randomized subjects with with EQ-5D analyzed.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 368 | 140
Participants
  mobility - Grade 1 | 129 | 39
  mobility - Grade 2 | 225 | 93
  mobility - Grade 3 | 11 | 5
  mobility - Missing | 3 | 3
  self-care - Grade 1 | 256 | 89
  self-care - Grade 2 | 102 | 46
  self-care - Grade 3 | 6 | 3
  self-care - Missing | 4 | 2
  usual activities - Grade 1 | 140 | 38
  usual activities - Grade 2 | 187 | 79
  usual activities - Grade 3 | 37 | 20
  usual activities - Missing | 4 | 3
  pain/discomfort - Grade 1 | 56 | 21
  pain/discomfort - Grade 2 | 270 | 95
  pain/discomfort - Grade 3 | 39 | 21
  pain/discomfort - Missing | 3 | 3
  anxiety/depression - Grade 1 | 195 | 64
  anxiety/depression - Grade 2 | 159 | 71
  anxiety/depression - Grade 3 | 10 | 2
  anxiety/depression - Missing | 4 | 3

40. Other Pre Specified Outcome: Number of Participants in the Euro Quality of Life (EQ-5D) Components for Mobility, Self-care, Usual Activities, Pain/Discomfort, and Anxiety/Depression at Follow-up Visit 8 (Week 139)
Description: The EQ-5D questionnaire was given to the subject at each visit. The EQ-5D questionnaire consisted of 5 ordinal categorical responses (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Number of participants with EQ-5D at follow-up visit 8, as measured by this questionnaire, was counted. The scores for the EQ-5D dimensions are assigned according to the level of problems reported (1 'no problems'; 2 'some problems'; 3 'extreme problems').
Time Frame: Follow-up Visit 8 (Week 139)
Population: The ITT population was all randomized subjects with with EQ-5D analyzed.
Measure: Number; unit: Participants
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo
Number analyzed (Participants) | 41 | 13
Participants
  mobility - Grade 1 | 9 | 2
  mobility - Grade 2 | 30 | 10
  mobility - Grade 3 | 1 | 1
  mobility - Missing | 1 | 0
  self-care - Grade 1 | 26 | 7
  self-care - Grade 2 | 12 | 3
  self-care - Grade 3 | 2 | 3
  self-care - MIssing | 1 | 0
  usual activities - Grade 1 | 13 | 2
  usual activities - Grade 2 | 19 | 7
  usual activities - Grade 3 | 8 | 4
  usual activities - Missing | 1 | 0
  pain/discomfort - Grade 1 | 5 | 1
  pain/discomfort - Grade 2 | 32 | 11
  pain/discomfort - Grade 3 | 3 | 1
  pain/discomfort - Missing | 1 | 0
  anxiety/depression - Grade 1 | 24 | 6
  anxiety/depression - Grade 2 | 15 | 7
  anxiety/depression - Grade 3 | 1 | 0
  anxiety/depression - Missing | 1 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs (TEAEs) data were collected after the first injection of study treatment and within 12 weeks after the last injection of study treatment.
Groups:
- Radium-223 Dichloride (Xofigo, BAY88-8223): Subjects received BSoC plus radium-223 50 kBq/kg body weight for 6 IV administrations separated by 4 weeks intervals.
- Placebo: Participants received BSoC plus isotonic saline for 6 IV administrations separated by 4 weeks intervals in double-blind phase.
- Placebo Randomized, Then Switched to Radium-223 Dichloride: Participants received BSoC plus isotonic saline for 6 IV administrations separated by 4 weeks intervals in double-blind phase; Participants received radium223 50 kBq/kg body weight for 6 intravenous administrations separated by 4 weeks intervals after unblinding to the end of study.
Arm/Group | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo | Placebo Randomized, Then Switched to Radium-223 Dichloride
Serious Adverse Events (participants affected / at risk) | 286 | 185 | 17
Other Adverse Events (participants affected / at risk) | 524 | 254 | 23
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo | Placebo Randomized, Then Switched to Radium-223 Dichloride
Anaemia (Blood and lymphatic system disorders) | 50/600 (70) | 25/301 (35) | 1/24 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Leukopenia (Blood and lymphatic system disorders) | 3/600 (3) | 0/301 (0) | 0/24 (0)
Neutropenia (Blood and lymphatic system disorders) | 3/600 (3) | 1/301 (1) | 0/24 (0)
Pancytopenia (Blood and lymphatic system disorders) | 5/600 (6) | 0/301 (0) | 1/24 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 14/600 (14) | 3/301 (3) | 1/24 (1)
Bone marrow failure (Blood and lymphatic system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Acute myocardial infarction (Cardiac disorders) | 1/600 (1) | 3/301 (3) | 0/24 (0)
Angina pectoris (Cardiac disorders) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Arrhythmia (Cardiac disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Atrial fibrillation (Cardiac disorders) | 3/600 (3) | 4/301 (4) | 0/24 (0)
Atrial flutter (Cardiac disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Atrioventricular block complete (Cardiac disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Cardiac arrest (Cardiac disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Cardiac failure (Cardiac disorders) | 2/600 (2) | 4/301 (4) | 0/24 (0)
Cardiac failure congestive (Cardiac disorders) | 4/600 (4) | 2/301 (2) | 0/24 (0)
Coronary artery disease (Cardiac disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Left ventricular failure (Cardiac disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Myocardial infarction (Cardiac disorders) | 3/600 (3) | 3/301 (3) | 0/24 (0)
Myocardial ischaemia (Cardiac disorders) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Supraventricular tachycardia (Cardiac disorders) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Left ventricular dysfunction (Cardiac disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Cardiopulmonary failure (Cardiac disorders) | 1/600 (1) | 2/301 (2) | 0/24 (0)
Acute coronary syndrome (Cardiac disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Cataract (Eye disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Glaucoma (Eye disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Abdominal distension (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Abdominal pain (Gastrointestinal disorders) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Ascites (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Constipation (Gastrointestinal disorders) | 8/600 (8) | 4/301 (4) | 0/24 (0)
Diarrhoea (Gastrointestinal disorders) | 3/600 (4) | 4/301 (4) | 0/24 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Dysphagia (Gastrointestinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Faecal incontinence (Gastrointestinal disorders) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Food poisoning (Gastrointestinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Gastritis (Gastrointestinal disorders) | 2/600 (2) | 1/301 (1) | 0/24 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Haematemesis (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Intestinal obstruction (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Intestinal perforation (Gastrointestinal disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Large intestine perforation (Gastrointestinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Mouth haemorrhage (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Nausea (Gastrointestinal disorders) | 9/600 (10) | 5/301 (6) | 0/24 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1/600 (1) | 1/301 (1) | 1/24 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Vomiting (Gastrointestinal disorders) | 11/600 (20) | 7/301 (7) | 0/24 (0)
Subileus (Gastrointestinal disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Erosive duodenitis (Gastrointestinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Asthenia (General disorders) | 3/600 (3) | 1/301 (1) | 0/24 (0)
Chest pain (General disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Death (General disorders) | 4/600 (4) | 1/301 (1) | 0/24 (0)
Fatigue (General disorders) | 6/600 (7) | 9/301 (9) | 0/24 (0)
Gait disturbance (General disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Malaise (General disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Mucosal inflammation (General disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Multi-organ failure (General disorders) | 3/600 (3) | 0/301 (0) | 0/24 (0)
Oedema (General disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Oedema peripheral (General disorders) | 4/600 (5) | 2/301 (2) | 0/24 (0)
Pyrexia (General disorders) | 6/600 (9) | 6/301 (7) | 0/24 (0)
Sudden death (General disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
General physical health deterioration (General disorders) | 15/600 (15) | 8/301 (8) | 1/24 (1)
Drug intolerance (General disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Cholecystitis (Hepatobiliary disorders) | 0/600 (0) | 0/301 (0) | 1/24 (1)
Cholestasis (Hepatobiliary disorders) | 1/600 (3) | 0/301 (0) | 0/24 (0)
Hepatic failure (Hepatobiliary disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Bile duct obstruction (Hepatobiliary disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Bronchitis (Infections and infestations) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Bronchopneumonia (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Catheter related infection (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Cellulitis (Infections and infestations) | 3/600 (3) | 1/301 (1) | 0/24 (0)
Clostridium difficile colitis (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Cystitis (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Gastroenteritis (Infections and infestations) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Herpes zoster (Infections and infestations) | 2/600 (2) | 1/301 (1) | 0/24 (0)
Infection (Infections and infestations) | 10/600 (12) | 3/301 (3) | 0/24 (0)
Listeriosis (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Lobar pneumonia (Infections and infestations) | 0/600 (0) | 2/301 (2) | 0/24 (0)
Lower respiratory tract infection (Infections and infestations) | 8/600 (9) | 2/301 (2) | 0/24 (0)
Oral candidiasis (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Pneumonia (Infections and infestations) | 17/600 (18) | 7/301 (8) | 1/24 (1)
Pneumonia primary atypical (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Postoperative wound infection (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Pyelonephritis (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Pyonephrosis (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Sepsis (Infections and infestations) | 7/600 (7) | 4/301 (4) | 0/24 (0)
Upper respiratory tract infection (Infections and infestations) | 1/600 (1) | 0/301 (0) | 1/24 (1)
Urinary tract infection (Infections and infestations) | 5/600 (5) | 6/301 (6) | 0/24 (0)
Urosepsis (Infections and infestations) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Abscess jaw (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Bacterial sepsis (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Staphylococcal infection (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Bursitis infective (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Lung infection (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Peritonitis bacterial (Infections and infestations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Device related infection (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Post procedural infection (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Gastroenteritis norovirus (Infections and infestations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Concussion (Injury, poisoning and procedural complications) | 0/600 (0) | 0/301 (0) | 1/24 (1)
Cystitis radiation (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Fall (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1/600 (1) | 1/301 (1) | 1/24 (1)
Hip fracture (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Injury (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Intentional overdose (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Patella fracture (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Sternal fracture (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Stent occlusion (Injury, poisoning and procedural complications) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Medical device complication (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 1/24 (1)
Skin laceration (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Device dislocation (Injury, poisoning and procedural complications) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Procedural pain (Injury, poisoning and procedural complications) | 2/600 (2) | 1/301 (1) | 0/24 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Aspartate aminotransferase increased (Investigations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Liver function test abnormal (Investigations) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Prostatic specific antigen increased (Investigations) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Anorexia (Metabolism and nutrition disorders) | 5/600 (5) | 1/301 (1) | 0/24 (0)
Cachexia (Metabolism and nutrition disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Dehydration (Metabolism and nutrition disorders) | 12/600 (20) | 3/301 (3) | 0/24 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 3/600 (3) | 1/301 (1) | 0/24 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Malnutrition (Metabolism and nutrition disorders) | 0/600 (0) | 0/301 (0) | 1/24 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0/600 (0) | 0/301 (0) | 1/24 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 61/600 (76) | 50/301 (56) | 1/24 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5/600 (8) | 2/301 (2) | 0/24 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0/600 (0) | 2/301 (2) | 0/24 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 14/600 (14) | 11/301 (11) | 1/24 (1)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Mobility decreased (Musculoskeletal and connective tissue disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1/600 (3) | 0/301 (0) | 1/24 (1)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Benign neoplasm of bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4/600 (4) | 0/301 (0) | 0/24 (0)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Bone marrow tumour cell infiltration (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 65/600 (67) | 38/301 (42) | 2/24 (2)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1/600 (2) | 0/301 (0) | 0/24 (0)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5/600 (5) | 2/301 (2) | 0/24 (0)
Benign urinary tract neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Aphasia (Nervous system disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Cerebral haemorrhage (Nervous system disorders) | 3/600 (3) | 2/301 (2) | 0/24 (0)
Cerebral ischaemia (Nervous system disorders) | 1/600 (1) | 3/301 (3) | 0/24 (0)
Cerebrovascular accident (Nervous system disorders) | 3/600 (3) | 0/301 (0) | 0/24 (0)
Convulsion (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Dementia (Nervous system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Dementia Alzheimer's type (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Dizziness (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Dysarthria (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Epilepsy (Nervous system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Facial palsy (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Haemorrhage intracranial (Nervous system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Hydrocephalus (Nervous system disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Monoparesis (Nervous system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Neuralgia (Nervous system disorders) | 0/600 (0) | 2/301 (3) | 0/24 (0)
Paraesthesia (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Paraparesis (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Paraplegia (Nervous system disorders) | 0/600 (0) | 2/301 (2) | 0/24 (0)
Peripheral motor neuropathy (Nervous system disorders) | 1/600 (1) | 3/301 (3) | 0/24 (0)
Polyneuropathy (Nervous system disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Somnolence (Nervous system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Spinal cord compression (Nervous system disorders) | 21/600 (21) | 16/301 (16) | 1/24 (1)
Syncope (Nervous system disorders) | 2/600 (2) | 1/301 (1) | 1/24 (1)
Transient ischaemic attack (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Tremor (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Brain oedema (Nervous system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Radicular syndrome (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Ischaemic stroke (Nervous system disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Nerve root compression (Nervous system disorders) | 4/600 (4) | 0/301 (0) | 0/24 (0)
Paresis cranial nerve (Nervous system disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Aggression (Psychiatric disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Confusional state (Psychiatric disorders) | 6/600 (6) | 3/301 (3) | 0/24 (0)
Depression (Psychiatric disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Intentional self-injury (Psychiatric disorders) | 1/600 (2) | 0/301 (0) | 0/24 (0)
Suicide attempt (Psychiatric disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Acute prerenal failure (Renal and urinary disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Calculus ureteric (Renal and urinary disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Haematuria (Renal and urinary disorders) | 11/600 (13) | 7/301 (9) | 0/24 (0)
Hydronephrosis (Renal and urinary disorders) | 8/600 (10) | 2/301 (2) | 0/24 (0)
Micturition urgency (Renal and urinary disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Renal failure (Renal and urinary disorders) | 7/600 (7) | 2/301 (2) | 0/24 (0)
Renal failure acute (Renal and urinary disorders) | 4/600 (4) | 0/301 (0) | 0/24 (0)
Renal pain (Renal and urinary disorders) | 0/600 (0) | 0/301 (0) | 1/24 (1)
Renal tubular necrosis (Renal and urinary disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Urinary bladder haemorrhage (Renal and urinary disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Urinary incontinence (Renal and urinary disorders) | 2/600 (2) | 0/301 (0) | 0/24 (0)
Urinary retention (Renal and urinary disorders) | 10/600 (10) | 9/301 (9) | 0/24 (0)
Haemorrhage urinary tract (Renal and urinary disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Prostatic haemorrhage (Reproductive system and breast disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0/600 (0) | 0/301 (0) | 1/24 (1)
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/600 (1) | 3/301 (4) | 0/24 (0)
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6/600 (6) | 5/301 (5) | 0/24 (0)
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4/600 (8) | 3/301 (3) | 0/24 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 7/600 (7) | 6/301 (6) | 0/24 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1/600 (1) | 1/301 (1) | 0/24 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/600 (0) | 2/301 (2) | 0/24 (0)
Circulatory collapse (Vascular disorders) | 1/600 (1) | 0/301 (0) | 0/24 (0)
Orthostatic hypotension (Vascular disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Peripheral ischaemia (Vascular disorders) | 0/600 (0) | 0/301 (0) | 1/24 (1)
Venous thrombosis (Vascular disorders) | 0/600 (0) | 1/301 (1) | 0/24 (0)
Deep vein thrombosis (Vascular disorders) | 4/600 (5) | 0/301 (0) | 0/24 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Radium-223 Dichloride (Xofigo, BAY88-8223) | Placebo | Placebo Randomized, Then Switched to Radium-223 Dichloride
Anaemia (Blood and lymphatic system disorders) | 161/600 (247) | 81/301 (104) | 8/24 (10)
Neutropenia (Blood and lymphatic system disorders) | 28/600 (37) | 3/301 (4) | 2/24 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 59/600 (71) | 15/301 (16) | 2/24 (2)
Abdominal pain (Gastrointestinal disorders) | 21/600 (21) | 13/301 (15) | 2/24 (2)
Constipation (Gastrointestinal disorders) | 105/600 (111) | 60/301 (68) | 2/24 (2)
Diarrhoea (Gastrointestinal disorders) | 153/600 (242) | 43/301 (60) | 7/24 (12)
Nausea (Gastrointestinal disorders) | 210/600 (294) | 98/301 (126) | 11/24 (12)
Vomiting (Gastrointestinal disorders) | 108/600 (151) | 34/301 (45) | 3/24 (3)
Asthenia (General disorders) | 35/600 (43) | 17/301 (19) | 2/24 (2)
Fatigue (General disorders) | 157/600 (192) | 73/301 (86) | 9/24 (10)
Oedema peripheral (General disorders) | 76/600 (82) | 29/301 (34) | 2/24 (2)
Pyrexia (General disorders) | 38/600 (58) | 15/301 (24) | 0/24 (0)
Nasopharyngitis (Infections and infestations) | 13/600 (13) | 8/301 (11) | 4/24 (4)
Urinary tract infection (Infections and infestations) | 47/600 (55) | 22/301 (23) | 5/24 (8)
Contusion (Injury, poisoning and procedural complications) | 12/600 (13) | 4/301 (4) | 3/24 (3)
Weight decreased (Investigations) | 74/600 (74) | 44/301 (45) | 2/24 (2)
Anorexia (Metabolism and nutrition disorders) | 104/600 (115) | 53/301 (57) | 4/24 (5)
Hypokalaemia (Metabolism and nutrition disorders) | 14/600 (16) | 6/301 (7) | 2/24 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2/600 (2) | 2/301 (2) | 3/24 (3)
Decreased appetite (Metabolism and nutrition disorders) | 36/600 (39) | 13/301 (13) | 1/24 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 287/600 (476) | 174/301 (321) | 11/24 (19)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2/600 (2) | 3/301 (3) | 2/24 (2)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 8/600 (8) | 15/301 (18) | 2/24 (2)
Dizziness (Nervous system disorders) | 45/600 (53) | 26/301 (30) | 2/24 (2)
Headache (Nervous system disorders) | 25/600 (29) | 9/301 (9) | 2/24 (2)
Paraesthesia (Nervous system disorders) | 16/600 (16) | 4/301 (4) | 2/24 (2)
Insomnia (Psychiatric disorders) | 31/600 (33) | 17/301 (17) | 0/24 (0)
Pollakiuria (Renal and urinary disorders) | 14/600 (15) | 5/301 (6) | 2/24 (2)
Urinary retention (Renal and urinary disorders) | 20/600 (20) | 12/301 (13) | 3/24 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 47/600 (54) | 21/301 (22) | 0/24 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No PI may disclose or publish information from the trial before publication of the principal and first communication arising from the trial, unless 12 months has elapsed after completion of the trial. There is restriction on the PI that the sponsor can review results communication prior to public release and can embargo regarding trial results for a period that is less/or equal to 60 days from the time submitted to the sponsor for review. Sponsor cannot require changes or extend the embargo.